CLINICAL TRIAL: NCT00433628
Title: Accuracy of Hemoglobin A1C to Predict Glycemia in HIV
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070094; 07-I-0094
Record Dates: First submitted 2007-02-09; First posted 2007-02-12 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-08-25

CONDITIONS: HIV; Diabetes; Hyperglycemia
Keywords: Hemoglobin A1C; HIV; Diabetes; Diabetes Type 2; Hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus; Hyperglycemia; Diabetes Mellitus, Type 2

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will see if HbA1C, the usual blood test for monitoring blood sugar control in diabetic patients, is as accurate in diabetic patients who also have HIV and will evaluate if alternative methods for monitoring blood sugar are preferred for HIV infected patients.

HIV-infected patients 18 years of age and older with type 2 diabetes or high blood sugar may be eligible for this study. Participants have two clinic visits (1 to 4 weeks apart) at the NIH Clinical Center. At the first visit they provide a detailed medical, social and family history and have blood and urine samples collected. Previous blood sugar values are also recorded. At the second visit, scheduled for 1 to 4 weeks after the first visit, blood and urine samples are collected. Some of the urine and blood samples are stored for future research on diabetes, HIV or related conditions.

...

DETAILED DESCRIPTION:
Diabetes mellitus is increasingly recognized among patients living with human immunodeficiency virus (HIV) infection. At present, there are no unique guidelines for the management of diabetes in patients with HIV. Diabetes in this population is managed in accordance with national guidelines for the management of diabetes in any patient. However, there have been small studies suggesting that hemoglobin A1C (HbA1C) may not be indicative of true glycemic control in HIV positive patients. There are currently no published prospective studies examining the ability of HbA1C to reflect glycemic control in HIV positive patients with diabetes. Since the incidence of HIV positive patients with lipodystrophy, glucose intolerance, and diabetes is steadily increasing with the widespread use of highly active antiretroviral therapy (HAART), the question of how best to monitor hyperglycemia in these patients is an important one.

This study, a prospective cross-sectional study of 100 patients, seeks to collect preliminary data to determine if HbA1C is appropriately reflecting plasma glucose in HIV positive patients. Patients with HIV and diabetes or hyperglycemia will have a fasting and a random plasma glucose and HbA1C collected as in normal diabetes patient care. They will also have two validated alternate markers of glycemic control drawn, fructosamine and Glycomark [R], to determine how well these markers may reflect actual glycemia. Fructosamine represents a measure of protein glycosylation whereas Glycomark [R] is a monosaccharide in plasma competitively inhibited in the renal tubules by glucose that reflects day-to-day hyperglycemia. In addition, hemolysis will be assessed to investigate this as one potential mechanism for why HbA1C may be a less accurate representation of glycemia in these patients. The determination of the value of HbA1C as a marker of glycemia in HIV positive patients with diabetes will assist with the monitoring and the management of this unique population with diabetes. The measurement of other glycemic markers may provide evidence towards potential superior markers of glycemia in these patients, and the study will provide insight into the possible mechanism of the HbA1C discrepancy.

ELIGIBILITY:
* INCLUSION CRITERIA:

Documented + HIV ELISA.

Diabetes mellitus (DM) will be defined as:

Documented diagnosis of type 2 diabetes mellitus or FPG greater than or equal to 126 mg/dl on two occasions or casual blood glucose greater than or equal to 200 mg/dL and symptoms of diabetes.

Impaired Fasting Glucose (IFG) defined as:

FPG greater than or equal to 100 mg/dl and less than 126 mg/dl on one or more occasions within past year.

Age 18+, male or female.

EXCLUSION CRITERIA:

Type 1 Diabetes.

Known current pregnancy or pregnancy within 6 mo.

Documented hemoglobinopathy.

Changes in antiretroviral therapy within 3 months.

History of anemia (Hb less than 9g/dL in past 6 months).

Active opportunistic Infection or opportunistic Infection within 3 mo.

Creatine greater than 1.8 mg/dL or known end stage renal disease (ESRD).

Changes in diabetes therapies within 3 mo (excluding dose adjustments).

Subject is deemed unable to comply with requirements of study participation.

Use of oral corticosteroid within the past 3 mo (stable dose inhaled steroids will be allowed).

Blood transfusion within 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175
Dates: Start 2007-02-07; Primary Completion 2008-11-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Washington Hospital Center, Washington D.C., District of Columbia
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland